CLINICAL TRIAL: NCT01103752
Title: Postoperative Cognitive Dysfunction After Total Knee or Hip Replacement Surgery in Fast-track Set-up
Status: Completed | Type: Observational
Sponsor: Lene Krenk (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Sponsor-Investigator, Lene Krenk, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-3-2009-096
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgery: This group (n=220) consist of patients undergoing hip or knee replacement in a fast-track setup and they are tested 3 times for postoperative cognitive dysfunction.
  Interventions: Other: no intervention, descriptive study

INTERVENTIONS:
Other: no intervention, descriptive study — no intervention, descriptive study

SUMMARY:
The aim of this study is to quantify the incidence of postoperative cognitive dysfunction in the elderly patient (>60y) after total hip or knee replacement surgery. The hypothesis is that the fast-track methodology with a mean hospital stay less than 3 days will help to minimize this reduction in memory and concentration.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or above
* ASA classification 1-4
* undergoing fast-track hip or knee replacement

Exclusion Criteria:

* anaesthesia within the past 90 days
* daily consumption of sleep or anxiety medication
* more than 35 units of alcohol per week
* lack of proper verbal and reading skills, Danish
* Serious hearing or visual impairment
* Mini mental status evaluation (MMSE) < 24
* Parkinsons Disease or other neurological disease causing functional impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing fast-track knee or hip replacement surgery at one of the hospitals participating (Hidovre, Holstebro, Hørsholm, Århus)
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lene Krenk, Doctor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- The Lundbeck Centre for fast-track hip/knee surgery, Copenhagen, Denmark